CLINICAL TRIAL: NCT02294149
Title: A Randomized Controlled Trial of Mammalian Omega 3 With Vitamin D3 in Patients at Risk of Chemotherapy Induced Peripheral Neuropathy.
Brief Title: Vit D3 and Omega 3 in Chemo Induced Neuropathy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Nathaniel Bouganim, Dr. Nathaniel Bouganim, Medical Oncologist at Royal Victoria Hospital muhc, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4086
Record Dates: First submitted 2014-11-17; First posted 2014-11-19 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Cancer; Neuropathy
Keywords: chemotherapy; Omega 3
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): A ineffective placebo drug with the same taste, route of administration and physical appearance as the study drug (omega 3/Vit D 3) that has received approval by health Canada.
  Interventions: Drug: placebo
- Omega 3 FA/Vitamin D3 sublingual (Experimental): patients will be allocated randomly to receive Sub-lingual Omega 3 FA and Vitamin D3 supplements for 6 months, twice daily ,1/2 tea spoon with instructions to keep it under the tongue for 45 sec.
  Interventions: Drug: mammalian Omega 3 Fatty acids

INTERVENTIONS:
Drug: mammalian Omega 3 Fatty acids — A mammalian oil derived Omega 3 FA that is a further concentrated and purified supplement as compared to the regular fish oil derived Omega 3 FA supplement.
  Arms: Omega 3 FA/Vitamin D3 sublingual
Drug: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether administration of mammalian Omega 3 FA(fatty acid) with Vitamin D3 supplements would lower or prevent the risk of neuropathy due to chemotherapy.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the impact of mammalian oil Omega 3 FA with Vitamin D3 supplementation on resolution or prevention of Taxanes or Platinum induced peripheral neuropathy compared with placebo. Patients will be allocated to receive the Omega 3 FA & Vitamin D3 supplements or placebo for 6 months. Approximately 600 patients in total will be enrolled in the 2 study arms. The evaluation of neuropathy will be accomplished by electromyography (EMG), Total neuropathy score(TNS), Brief pain inventory (BFI) and the 11-item FACT/GOG-Ntx, version 4 questionnaire (a subscale validated to assess neuropathy due to chemotherapy). In addition, other validated functional measures such as "Time to button a six hole shirt" and "50 ft walk speed test" will be used to test patients physical limitations imposed by peripheral neuropathy. All our patients will undergo an EMG at their first visit, in 3 months and after 6months. Previously mentioned functional measures will also be completed at the patients' first visit, in 3 months and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Will be receiving chemotherapy(Platinums and/or Taxanes) in the following 2 weeks.
* Histologically confirmed diagnosis of cancer
* ECOG 0 to 2

Exclusion Criteria:

* Prior chemotherapy treatment
* Pre-existing peripheral PN due to DM,HIV, alcohol abuse, thyroid dysfunction and hereditary PN associated disorders.
* Taking any nutritional supplement( fish oil, vitamins and minerals) at least there months before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
percentage of participants with a 50% decreases in Total neuropathy score | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- McGill university health center, Royal Victoria hospital, Montreal, Quebec, Canada